CLINICAL TRIAL: NCT04837352
Title: Obstacles and Levers of the Therapeutic Adherence of Multiple Sclerosis Patients
Brief Title: Therapeutic Adherence of Multiple Sclerosis Patients
Acronym: FELSA-SEP
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P00105
Record Dates: First submitted 2021-02-02; First posted 2021-04-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Theory of Planned Behaviour; Therapeutic adherence; Sociocognitive and interpersonal factors
MeSH Terms: conditions — Multiple Sclerosis; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis patients: Patients with multiple sclerosis over 18 years old who have already started a long-term treatment and consent to participate to the study
  Interventions: Other: Study of the role of sociocognitive factors

INTERVENTIONS:
Other: Study of the role of sociocognitive factors — Questionnaires

SUMMARY:
The goal of this study is to assess the role of sociocognitive and interpersonal factors in the therapeutic adherence of multiple sclerosis patients. This study will provide a better understanding of the socio-psychological issues associated with different types of non-adherence to treatment, and identify the risk factors and vulnerability of each patient.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic and progressive disease that affects young adults (between 20 and 40 years old), impacting significantly the patients quality of life.

The adherence to therapy affects the long-term functional clinical course (lower risk of relapses, reduction in disability progression and quality of life). The non-adherence rate to therapy in multiple sclerosis is estimated at 40%. The main identified causes of non-adherence are: forgetting to take treatment and adverse effects of drugs.

Sociocognitive models as the Theory of Planned Behaviour (TPB) have been developed to help to understand and predict health-related behaviours. This model postulates that the intention to adopt a behaviour is one of the major determinants in the context of health. This intention comes from three independent elements :

* Personal positive or negative attitudes towards the behaviour,
* Social expectations or entourage perception (subjective norms),
* Difficulty in accomplishing this behaviour (perceived control)

Multiple sclerosis adherence to therapy studies have mainly focused on somatic variables (physical disability, illness duration, type of treatment) and some clinical variables (cognitive impairment, fatigue, depression). The few studies that have examined the multiple sclerosis therapeutic adherence determinants have mainly taken a one-dimensional perspective, such as perceived control.

In the FELSA-SEP study, the role of sociocognitive factors (norms and beliefs, perceived threat to disease and health behaviours) and interpersonal factors (social support, patient-doctor relationship) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis defined according to McDonald criteria;
* Already undergone or beginning substantive treatment (self-managed, excluding treatment administered in hospital)
* Aged ≥ 18 years;
* Given the informed consent form.

Exclusion Criteria:

* Severe cognitive impairment (score below the 5th percentile);
* Any associated neurological pathology or serious or chronic somatic disease (cancer);
* Being under a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with multiple sclerosis who will be recruited during a routine neurological consultation and who present eligibility criterion.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence evaluated by a Likert scale | 6 months
  This 19-item self-questionnaire provides 5 sub-scores corresponding to each of the sub-dimensions (Attitudes, Subjective norms, Perception of control, Behavioural intention and Behaviour) and an overall score (sum of the 5 sub-scores).

SECONDARY OUTCOMES:
Perceived threat measured with a self-assessment form | 3 weeks
  The perceived threat will be measured with a self-assessment form using a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). This 11-item self-questionnaire provides 2 sub-scores and an overall score (sum of the 2 sub-scores).
Perceived interpersonal relationships quality measure by the perceived social support questionnaire (QSSP) | 6 months
  * The QSSP is a 6 items questionnaire which assess availability and satisfaction with respect to perceived social support.
  * 4-Point ordinal Alliance Scale (11-items 4-PAS). This self-questionnaire concerns the patient's perception about the therapeutic alliance.
Perceived interpersonal relationships quality measure by the 4-Point ordinal Alliance Scale (11-items 4-PAS) | 6 months
  The 4-Point ordinal Alliance Scale (11-items 4-PAS). This self-questionnaire concerns the patient's feelings about the therapeutic alliance and includes eleven items, placing the patient on 5-point scale on : the patient's feeling about the doctor's ability to help him/her; his/her understanding of the symptoms of the illness; the psychological improvement felt; the adaptation to the doctor-patient relationship; the doctor's availability and competence; the clarity of the information given by the doctor and the understanding he/she shows; the doctor's desire of clinical improvement; the quality of the relationship and the understanding of psychological difficulties
Illness duration in days | 3 weeks
  In order to evaluate the vulnerability and protective factors related to somatic disease illness duration will be evaluated.
Handicap will be evaluated by the Expanded Disability Status Scale (EDSS) | 3 weeks
  In order to evaluate the vulnerability and protective factors related to somatic the handicap will be evaluated by the EDSS. The EDSS quantifies disability in eight Functional Systems (FS) by assigning a Functional System Score in each of these functional systems.
  The clinical meaning of each possible result goes from 0.0: Normal Neurological Exam to 10.0: Death
Relapses number | 3 weeks
  In order to evaluate the vulnerability and protective factors related to somatic disease number of relapses will be evaluated
Fatigue perceived through the FSS (Fatigue Severity Scale) | 3 weeks
  In order to evaluate the vulnerability and protective factors related to somatic disease fatigue will be evaluated. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Cognitive disorders through the SDMT (Symbol Digit Modalities Test) | 3 weeks
  In order to evaluate the vulnerability and protective factors related to somatic disease cognitive disorders will be evaluated The SDMT is a sign coding test that assesses attentional abilities (sustained attention and speed of processing information). Participants are required to use a coded key to match nine abstract symbols paired with numerical digits. The final score is the correct number of substitutions in 90 seconds, and scores range between 0 and 110.
Anxiety-depressive symptoms measured by the Hospital Anxiety and Depression Scale (HADS) | 3 weeks
  The vulnerability and protective factors linked to psychological functioning- as Anxiety-depressive symptoms will be determined.
  - Personality traits: Big Five Inventory-FR questionnaire (BFI-FR)
Personality traits measured by the Big Five Inventory-FR questionnaire (BFI-FR) | 3 weeks
  The vulnerability and protective factors linked to psychological functioning as personality traits will be determined.
  The Big Five personality traits is a suggested grouping for personality traits. The theory identifies five factors:
  * openness to experience (inventive/curious vs. consistent/cautious)
  * conscientiousness (efficient/organized vs. extravagant/careless)
  * extraversion (outgoing/energetic vs. solitary/reserved)
  * agreeableness (friendly/compassionate vs. challenging/callous)
  * neuroticism (sensitive/nervous vs. resilient/confident)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lenne, Principal Investigator — Hôpital Saint Vincent de Paul, Lille
Locations (4):
- France (4):
  - CHRU DE Bordeaux, Bordeaux
  - Hôpital Saint-Vincent de Paul, Lille
  - Hôpital Saint-Philibert, Lomme
  - CHRU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No